CLINICAL TRIAL: NCT02277249
Title: Transvaginal Versus Transabdominal Digoxin Prior to Second-trimester Abortion: a Pilot Study of Patient Preference
Brief Title: Transvaginal Versus Transabdominal Digoxin Prior to Second-trimester Abortion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: IRB#12-001241
Record Dates: First submitted 2014-10-21; First posted 2014-10-28 (Estimated); Results first posted 2016-10-19 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2016-11

CONDITIONS: Abortion, Induced
MeSH Terms: interventions — Digoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transvaginal digoxin (Other): Transvaginal administration of digoxin for inducing fetal death prior to second-trimester abortion
  Interventions: Drug: Digoxin (transvaginal administration)
- Transabdominal digoxin (Other): Transabdominal administration of digoxin for inducing fetal death prior to second-trimester abortion
  Interventions: Drug: Digoxin (transabdominal administration)

INTERVENTIONS:
Drug: Digoxin (transvaginal administration) — Transvaginal digoxin administration prior to second-trimester abortion. This is only listed as a "Procedure/Surgery" type intervention because the mode of digoxin administration (transvaginal versus transabdominal) is what is being studied.
  Arms: Transvaginal digoxin
Drug: Digoxin (transabdominal administration) — Transabdominal digoxin administration prior to second-trimester abortion. This is only listed as a "Procedure/Surgery" type intervention because the mode of digoxin administration (transvaginal versus transabdominal) is what is being studied.
  Arms: Transabdominal digoxin

SUMMARY:
Current practice for the provision of late second trimester abortion (dilation and evacuation, or D&E) often involves the administration of digoxin into the fetal compartment to induce fetal demise prior to the procedure. Digoxin may be administered transabdominally or transvaginally into the fetal compartment. Both modes of administration have been shown in prospective studies to be highly effective and safe. Both modes of administration are considered standard of care. This pilot study will directly compare transabdominal and transvaginal digoxin with respect to patient preference (i.e, patient pain score describing discomfort with injection).

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* Singleton viable gestation
* Identifying as primarily English-speaking
* Body mass index less than 40 kilograms/meters squared
* Already a consented patient for second-trimester abortion procedure with digoxin to be performed for termination of pregnancy at the study site
* No medical contraindication to digoxin (i.e., no cardiac dysfunction, no renal dysfunction, no hypersensitivity to digoxin)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-10; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Transvaginal Digoxin | Transabdominal Digoxin
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Transvaginal Digoxin | Transabdominal Digoxin | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: Years] | 26.8 (6.7) | 26.6 (6.1) | 26.7 (6.4)
Gender [Count of Participants; unit: Participants]
  Female | 30 | 30 | 60
  Male | 0 | 0 | 0
Gestational Age [Mean (Standard Deviation); unit: Weeks] | 21.5 (1.2) | 21.4 (1.6) | 21.4 (1.4)
Parity [Mean (Standard Deviation); unit: Births] | 0.8 (0.8) | 0.87 (1.2) | 0.83 (1.0)
Body Mass Index [Mean (Standard Deviation); unit: Kilograms/meters squared] | 27.4 (5.0) | 26.7 (4.8) | 27.1 (4.8)

OUTCOME MEASURES:

1. Primary Outcome: Patient Discomfort With Digoxin Injection (Pain Score)
Description: Pain score (indicated by patient reporting pain level from 0 ("no hurt") to 5 ("hurts worst") at time of digoxin injection)
Time Frame: At time of study (immediate)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Transvaginal Digoxin | Transabdominal Digoxin
Number analyzed (Participants) | 30 | 30
Units on a scale | 2.21 (1.33) | 1.88 (1.54)
Statistical Analysis 1: Comparison: Transvaginal Digoxin vs Transabdominal Digoxin; No power calculation performed given that this was a pilot study. The null hypothesis was that there would be no difference in pain score with injection between the two study arms. The Wilcoxon rank sum test was selected because of the study's small sample size and the non-normal distribution of pain scores. Intention to treat analyses were used; Test type: Superiority or Other; p = 0.36, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Transvaginal Digoxin | Transabdominal Digoxin
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

LIMITATIONS AND CAVEATS:
There was crossover between treatment arms (4 subjects in the transvaginal group received transabdominal digoxin). This study is limited by its small sample size and attendant statistical power.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No